CLINICAL TRIAL: NCT03453684
Title: Preoperative Vancomycin Administration for Surgical Site Prophylaxis: Plasma and Soft Tissue Concentrations in Pediatric Neurosurgical and Orthopedic Patients
Brief Title: Pharmacokinetics of Preoperative Vancomycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1411
Record Dates: First submitted 2018-02-14; First posted 2018-03-05 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Surgical Site Infection; Vancomycin
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of Vancomycin (Experimental): Administration of Vancomycin 15 mg/kg over 1 hour prior to surgical incision
  Interventions: Drug: Administration of Vancomycin

INTERVENTIONS:
Drug: Administration of Vancomycin — Intravenous Vancomycin Administration
  Other Names: Vancomycin Hydrochloride

SUMMARY:
A study of plasma and tissue vancomycin pharmacokinetics in pediatric surgical patients.

DETAILED DESCRIPTION:
Background: Vancomycin is used for antibiotic prophylaxis in pediatric surgical patients without a complete understanding of plasma and soft tissue pharmacokinetics. Guidelines recommend incision within 60 minutes after administration; however, tissue concentrations of vancomycin at that early time may not be therapeutic. The Investigators conducted a study of plasma and tissue concentrations in pediatric neurosurgical and orthopedic patients to characterize intraoperative vancomycin pharmacokinetics.

Patients, ages (0.1-18.8 years), undergoing posterior spinal fusion (n=30) or ventriculoperitoneal shunt placement (n=30), received intravenous vancomycin 15 mg/kg over one hour. Skin biopsies were taken at incision and skin closure. Blood samples were also collected at incision and closure; additional samples were drawn at 2- and 4-hours if patient was still in surgery. Population pharmacokinetic (PK) analysis was performed to characterize PK parameter estimates and to develop a model of intraoperative plasma and tissue vancomycin concentrations vs. time.

ELIGIBILITY:
Inclusion Criteria:

1. Neurosurgery patients between the ages of 31 days up to 18 years
2. Receiving a single dose of vancomycin administered prior to surgery for cerebrospinal fluid (CSF) shunt placement or revision.
3. Orthopedic surgical patients between the ages of 31 days up to 18 years
4. Receiving a single dose of vancomycin administered prior to surgery for definitive spinal fusion.

Exclusion Criteria:

1. Patients already receiving vancomycin for treatment of an active infection,
2. Patients who have a Creatinine ≥1.2,
3. Patients who's creatinine clearance less than 50,
4. Known chronic renal failure and are on dialysis,
5. Patients with a known allergy to vancomycin, not including Red Man Syndrome.

Ages: 31 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2015-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Brooks-Peterson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients scheduled to undergo posterior spinal fusion 30 patients scheduled to undergo ventriculo-peritoneal (VP) shunt placement
Period: Overall Study
Arm/Group | Administration of Vancomycin
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Analysis: V˅c
Description: Volume of the central compartment. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: 1 Day (measured and combined from the time of the incision, through 2 hours after the incision, 4 hours after the incision, until when the incision is closed).
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L
  Typical value | 2.56
  w^2 | 1.14
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall SE of the estimate = 0.009 — Standard error of the estimate of Typical value: 0.45 Standard error of the estimate of w^2: 0.39

2. Primary Outcome: Pharmacokinetics Analysis: V˅2
Description: Volume of the peripheral compartment Typical value. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L/35kg
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L/35kg | 5.30
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall Standard Error of the Estimate = 9.85 — Standard error of the estimate of Typical value: 0.61 Standard error of the estimate of ꙍ^2 (intersubject variability): ^a (fixed to 0)

3. Primary Outcome: Pharmacokinetics Analysis: Q
Description: Intercompartmental clearance between central compartment (Vc) and peripheral compartment (V2) Typical Value. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L/min
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L/min | 0.12
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall Standard Error of the Estimate = 8.37 — Standard error of the estimate of Typical value: 0.02 Standard error of the estimate of ꙍ^2 (intersubject variability): ^a (fixed to 0)

4. Primary Outcome: Pharmacokinetics Analysis: Cle
Description: Elimination clearance. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L/min/1.73 m^2
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L/min/1.73 m^2
  Typical value | 0.09
  ꙍ^2 (Intersubject variability) | 0.13
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall Standard Error of the Estimate = 4.83 — Standard error of the estimate of Typical value: 0.003 Standard error of the estimate of ꙍ^2 (intersubject variability): 0.03

5. Primary Outcome: Pharmacokinetics Analysis: sf˅V2
Description: Scaling Factor for Body weight covariate for V2 (Volume of the peripheral compartment) Typical Value. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L/35kg
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L/35kg | 1.01
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall Standard Error of the Estimate = 17.21 — Standard error of the estimate of Typical value: 0.13

6. Primary Outcome: Pharmacokinetics Analysis: sf˅Cle
Description: Scaling Factor for Body weight covariate for Cle (elimination clearance) Typical Value. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: L/min/1.73m^2
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
L/min/1.73m^2 | 1.69
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; SE of the estimate of Typical Value = 0.20

7. Primary Outcome: Pharmacokinetics Analysis: K˅skin0
Description: Accounts for the equilibration rate between plasma and skin. Typical Value should be read as 3.6E-05. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: min^-1
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
min^-1
  Typical value | 3.6
  ꙍ^2 (Intersubject variability) | 2.0
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; SE of the estimate of Typical Value = 2.1 — Standard error of the estimate of Typical value should be read as: 2.1E-06 Standard error of the estimate of ꙍ^2 (intersubject variability): 0.24

8. Primary Outcome: Pharmacokinetics Analysis: PC
Description: Partition coefficient, models skin drug concentration between plasma and skin. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: Coefficient
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
Coefficient
  Typical value | 32.0
  ꙍ^2 (Intersubject variability) | 3.7
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; SE of the estimate of Typical Value = 2.3 — Standard error of the estimate of ꙍ^2 (intersubject variability): 0.08

9. Primary Outcome: Pharmacokinetics Analysis: δ ˅R-plasma
Description: Proportional or relative intrasubject variability for plasma data Typical Value. There is no unit of measure for this measurement. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: No unit of measure
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
No unit of measure | 0.23
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; Overall Standard Error of the Estimate = 10.80 — Standard error of the estimate of Typical value: 0.02

10. Primary Outcome: Pharmacokinetics Analysis: δ ˅A-skin
Description: Additive intrasubject variability for skin data Typical Value. This outcome measure was pre-specified to utilize advanced mathematical modeling for this assessment. No measure of central tendency is available.
Time Frame: as for outcome 1
Population: One participant was excluded because the sample was lost.
Measure: Number; unit: μg
Arm/Group | Administration of Vancomycin
Number analyzed (Participants) | 59
μg | 7.5
Statistical Analysis 1: Comparison: Administration of Vancomycin; Test type: Other; SE of the estimate of Typical Value = 0.90

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Administration of Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

LIMITATIONS AND CAVEATS:
Outcome measures were determined by complex mathematical modeling utilizing the pharmacokinetics estimates listed above. Outcome measures are described as necessary report the pharmacokinetic data. Outcome measures reflect the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes